CLINICAL TRIAL: NCT04335552
Title: Pragmatic Factorial Trial of Hydroxychloroquine, Azithromycin, or Both for Treatment of Severe SARS-CoV-2 Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment, strong evidence from larger trials of no therapeutic benefit
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PRO00105339
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Results first posted 2021-05-12 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV-2
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care; Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Intervention Model Description: Patients will be initially randomized to one of two arms in a 1:1 ratio: 1) Standard of care treatment or 2) Standard of care treatment plus 5 days of hydroxychloroquine. Participants who meet eligibility criteria to receive azithromycin will undergo a second randomization in a 1:1 ratio to receive additional concurrent therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard of care (Active Comparator)
  Interventions: Other: Standard of care
- Standard of care plus hydroxychloroquine (Experimental): Standard of care plus hydroxychloroquine for 5 days
  Interventions: Other: Standard of care; Drug: Hydroxychloroquine
- Standard of care plus azithromycin (Experimental): Standard of care plus azithromycin for 5 days
  Interventions: Other: Standard of care; Drug: Azithromycin
- Standard of care plus hydroxychloroquine plus azithromycin (Experimental): Standard of care plus hydroxychloroquine plus azithromycin for 5 days
  Interventions: Other: Standard of care; Drug: Hydroxychloroquine; Drug: Azithromycin

INTERVENTIONS:
Other: Standard of care — Standard of care
Drug: Hydroxychloroquine — Hydroxychloroquine will be administered orally or via feeding tube at a dosage of 800 mg on day 1, followed by 600 mg daily on days 2-5
  Arms: Standard of care plus hydroxychloroquine; Standard of care plus hydroxychloroquine plus azithromycin
Drug: Azithromycin — Azithromycin will be administered orally or via feeding tube at a dosage of 500 mg on day 1, followed by 250 mg daily on days 2-5
  Arms: Standard of care plus azithromycin; Standard of care plus hydroxychloroquine plus azithromycin

SUMMARY:
This is a pragmatic, randomized, open-label, incomplete factorial with nested randomization clinical trial evaluating the efficacy and safety of two potential treatments for hospitalized patients with confirmed SARS-CoV-2 infection. Participants who are hospitalized and have a positive nucleic acid amplification test for SARS-CoV-2 will undergo an initial randomization in a 1:1 ratio to one of the following regimens:

Arm 1: Standard of care alone

Arm 2: Standard of care plus hydroxychloroquine

Participants who meet eligibility criteria to receive azithromycin will undergo a second randomization in a 1:1 ratio to receive additional concurrent therapy. This will effectively result in four treatment groups:

1. Standard of care alone
2. Standard of care plus hydroxychloroquine
3. Standard of care plus azithromycin
4. Standard of care plus hydroxychloroquine plus azithromycin

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to participating hospital with symptoms suggestive of COVID-19 infection OR develop symptoms of COVID-19 during hospitalization
2. Subject (or legally authorized representative) can provide written informed consent (in English or Spanish) affirming intention to comply with planned study procedures prior to enrollment
3. Male or female adult aged 12 years or older at the time of enrollment
4. Has laboratory-confirmed SARS-CoV-2 infection determined by a validated nucleic acid amplification assay (public health or commercial) in any respiratory specimen collected within 14 days of randomization
5. Illness of any duration that includes

   * Radiographic evidence of pulmonary infiltrates (chest X-ray or CT scan) OR
   * Clinical documentation of lower respiratory symptoms (cough, shortness of breath, wheezing) OR
   * Any documented SpO2 ≤ 94% on room air OR
   * Any inpatient initiation or supplemental oxygen regardless of documented cause

Exclusion Criteria:

1. Participating in any other clinical trial of an experimental agent for COVID-19
2. On hydroxychloroquine at any time during hospitalization, or within 180 days of hospitalization for COVID-19 regardless of indication
3. History of G6PD deficiency, cirrhosis, long QT syndrome or porphyria of any classification
4. Most recent ECG prior to time of screening with QTc of ≥500 msec
5. Known hypersensitivity to hydroxychloroquine or 4-aminoquinoline derivatives
6. Death anticipated within 48 hours of enrollment
7. Inability to obtain informed consent from the patient or designated medical decision maker

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Stout, MD, Principal Investigator — Duke University Hospital
Locations (4):
- United States (4):
  - Duke Regional Hospital, Durham, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin
Started | 2 | 4 | 3 | 2
Completed | 1 | 4 | 3 | 2
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin | Total
Number analyzed (Participants) | 2 | 4 | 3 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (20.5) | 59.0 (14.1) | 57.0 (4.2) | 50.3 (12.5) | 54.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 3
  Male | 1 | 3 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 2 | 1 | 6
  Not Hispanic or Latino | 2 | 1 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 1 | 3 | 2 | 1 | 7
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 4 | 3 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization (WHO) Ordinal Scale Measured at 14 Days After Enrollment
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.
Time Frame: Day 14
Population: Intention to treat (includes all randomized, excludes 1 participant who withdrew prior to outcome measurement)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin
Number analyzed (Participants) | 1 | 4 | 3 | 2
units on a scale | 1 (NA) — Only one measurement | 2.5 (3) | 5.3 (3.8) | 4.5 (5.0)

2. Secondary Outcome: Number of Participants Who Died During the Index Hospitalization
Time Frame: Index hospitalization, up to 46 days
Population: Intention to treat (1 participant who withdrew not included)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin
Number analyzed (Participants) | 1 | 4 | 3 | 2
Participants | 0 | 1 | 2 | 1

3. Secondary Outcome: Number of Days on Mechanical Ventilation
Time Frame: Baseline
Population: Intention to treat (1 participant who withdrew excluded)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin
Number analyzed (Participants) | 1 | 4 | 3 | 2
days | 0 (NA) — Only 1 observation | 5.5 (11) | 8.67 (15) | 0 (0)

4. Secondary Outcome: Number of Patients Not Receiving Mechanical Ventilation at Baseline Who Progress to Requiring Mechanical Ventilation During the Index Hospitalization
Time Frame: Index hospitalization, up to 46 days
Population: Intention to treat excluding 1 participant who withdrew
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin
Number analyzed (Participants) | 1 | 4 | 3 | 2
Participants | 0 | 1 | 1 | 0

5. Secondary Outcome: WHO Ordinal Scale Measured at 28 Days After Enrollment
Description: as for outcome 1
Time Frame: Day 28
Population: Intention to treat excluding 1 participant who withdrew
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin
Number analyzed (Participants) | 1 | 4 | 3 | 2
score on a scale | 1 (NA) — Only 1 participant | 2.8 (3.5) | 5.3 (3.8) | 4.5 (5.0)

6. Secondary Outcome: Hospital Length of Stay in Days for the Index Hospitalization
Time Frame: Index hospitalization, up to 46 days
Population: Intention to treat excluding 1 participant who withdrew
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin
Number analyzed (Participants) | 1 | 4 | 3 | 2
days | 6 (NA) — Only 1 participant | 9 (11) | 14.7 (14.6) | 2.5 (0.7)

7. Secondary Outcome: Number of Participants With All-cause Study Medication Discontinuation
Description: Number of participants who discontinued study medication for any reason
Time Frame: Index hospitalization, up to 46 days
Population: Intention to treat excluding 1 participant who withdrew
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin
Number analyzed (Participants) | 1 | 4 | 3 | 2
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Severe Adverse Events
Time Frame: Day 14
Population: Intention to treat excluding 1 participant who withdrew
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin
Number analyzed (Participants) | 1 | 4 | 3 | 2
Participants | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Standard of Care | Standard of Care Plus Hydroxychloroquine | Standard of Care Plus Azithromycin | Standard of Care Plus Hydroxychloroquine Plus Azithromycin
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/4 | 2/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/4 | 1/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4 | 0/3 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=1) | Standard of Care Plus Hydroxychloroquine (N=4) | Standard of Care Plus Azithromycin (N=3) | Standard of Care Plus Hydroxychloroquine Plus Azithromycin (N=2)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Acute respiratory failure requiring intubation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT04335552/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT04335552/SAP_003.pdf
  • Informed Consent Form (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT04335552/ICF_002.pdf